CLINICAL TRIAL: NCT05922306
Title: A Multicenter, Prospective Cohort Study: Efficacy of NA Combined With PEG-IFN-α2b Continuous Versus Pulsed Therapy for 96 Weeks in Patients With Chronic Hepatitis B.
Brief Title: Efficacy of NA Combined With PEG-IFN-α2b in the Continuous Versus Pulsed Treatment of Patients With Chronic Hepatitis B
Acronym: EPCP
Status: Recruiting | Phase: Early Phase 1 | Type: Interventional
Sponsor: Anhui Medical University (Other)
Collaborators: The First Affiliated Hospital, University of Science and Technology of China (Other); The Second Hospital of Anhui Medical University (Other); Chaohu Hospital of Anhui Medical University (Other); The First Affiliated Hospital of Bengbu Medical University (Other)
Responsible Party: Principal Investigator, Yufeng Gao, Clinical Professor, Anhui Medical University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: LCYJ2021ZD006
Record Dates: First submitted 2023-06-02; First posted 2023-06-28 (Actual); Last update posted 2023-06-28 (Actual); Status verified 2023-06

CONDITIONS: Hepatitis B, Chronic
MeSH Terms: conditions — Hepatitis B, Chronic

STUDY DESIGN:
Masking Description: Participants and investigators will be informed of the treatment protocol. Participants will be grouped according to the random number method at initial entry and will be given the option to continue in the current cohort or withdraw from the cohort study at their own discretion after treatment assessment at each node.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Continuous Combination Therapy Cohort (Active Comparator): Patients with primary CHB with HBsAg ≥ 1500 IU/ml and HBV-DNA < 500 IU/ml and patients with CHB after treatment with NAs will be enrolled. After fully informed consent, pegylated interferon alpha-2b 180µg will be administered by subcutaneous injection once a week for up to 96 weeks.
  Interventions: Drug: PEGylated recombinant human interferon alpha-2b injection
- Pulsed Combination Therapy Cohort (Experimental): Patients with primary CHB with HBsAg ≥ 1500 IU/ml and HBV-DNA < 500 IU/ml and patients with CHB after treatment with NAs will be enrolled. After fully informed consent, pegylated interferon alpha-2b 180µg will be administered by subcutaneous injection once weekly for 8 weeks of treatment and discontinued for 4 weeks up to 96 weeks.
  Interventions: Drug: PEGylated recombinant human interferon alpha-2b injection

INTERVENTIONS:
Drug: PEGylated recombinant human interferon alpha-2b injection — Continuous combination therapy: pegylated interferon alpha-2b 180µg, subcutaneously once a week for 96 weeks, combined with NAs throughout the treatment period.
  Other Names: Nucleotide analogues
  Arms: Continuous Combination Therapy Cohort
Drug: PEGylated recombinant human interferon alpha-2b injection — Pulsed combination therapy: pegylated interferon alpha-2b 180µg once weekly by subcutaneous injection for 8 weeks with 4 weeks off for a total treatment duration of 96 weeks, combined with NAs throughout the treatment period.
  Other Names: Nucleotide analogues
  Arms: Pulsed Combination Therapy Cohort

SUMMARY:
Previous studies have shown that there are alterations in the number and affinity of interferon receptors during interferon therapy and that such alterations recover to varying degrees some time after the end of treatment. It can be conjectured that the rest period of pulsed therapy facilitates the recovery of type I interferon receptors and thus the next round of IFN therapy compared to a continuous regimen of interferon.

DETAILED DESCRIPTION:
A large-sample, multicenter, prospective, real-world study using NAs in combination with PEG-IFN-α-2b for the treatment of CHB patients with continuous or pulsed combination therapy over a course of up to 96 weeks is proposed to compare the differences in clinical cure rates and E antigen conversion rates between groups. Multiple novel markers of hepatitis B infection, including HBV pgRNA, HBcrAg and anti-HBcAb quantification, were dynamically measured at baseline, 12, 24, 48, 72 and 96 weeks to explore the appropriate strategy for achieving clinical cure rates in CHB patients treated with NAs in combination with PEG-IFN-α-2b.

ELIGIBILITY:
Inclusion Criteria:

1. Age 18 to 60 years, both sexes (both 18 and 60 years)
2. HBsAg positive for more than 6 months;
3. NAs treated patients on continuous NA therapy for more than 6 months with HBsAg ≥ 1500 IU/ml and HBV-DNA < 500 IU/ml at enrolment;
4. Primary treated patients with surface antigen >1500 IU, unlimited E antigen and unlimited HBV DNA at enrolment, meeting the treatment indications of the 2019 edition of the guidelines for the prevention and treatment of chronic hepatitis B.
5. negative urine or serum pregnancy test within 24 hours prior to the first dose (for women of childbearing age)

Exclusion Criteria:

1. Combined active hepatitis A, C, D, E and/or HIV infection;
2. Patients who are on future and intend to continue to use tibivudine
3. methaemoglobin greater than 100ng/ml at screening; or methaemoglobin that has not remained stable for 3 months prior to the trial and/or liver imaging suggestive of liver tumours;
4. decompensated liver disease (Child-Pugh score ≥ 7), meaning that patients will be excluded if one of the following is met: prolonged prothrombin time ≥ 3 seconds, serum bilirubin > 34umol/L, history of hepatic encephalopathy, history of oesophageal variceal bleeding, ascites;
5. pregnant or lactating women or patients with planned pregnancy during the study period and unwilling to use contraception
6. Neutrophil count < 1.5 x 10^9/L or platelet count < 90 x 10^9/L and creatinine > 1.5 ULN
7. History of severe psychiatric illness, especially depression. Major psychosis defined as major depressive disorder or psychosis, suicide attempts, hospitalisation for psychosis or incapacity for a period of time due to psychosis;
8. history of immune-mediated disease (e.g. inflammatory bowel disease, idiopathic thrombocytopenic purpura, lupus erythematosus, autoimmune haemolytic anaemia, scleroderma, severe psoriasis, rheumatoid arthritis) or abnormally elevated levels of autoimmune antibodies
9. Patients with severe combined diseases of the heart, lungs, kidneys, brain, blood and other vital organs, combined with other malignancies
10. History of severe epilepsy or current treatment with anti-epileptic drugs. Unstable control of diabetes mellitus, hypertension, thyroid disease, etc. Patients with a history of severe retinopathy or as indicated by other evidence of retinopathy;
11. History of any organ transplantation and existing functional grafts (except corneal or hair transplants);
12. Patients who are allergic to interferon and its drug components and who, in the judgment of the investigator, are unsuitable for interferon application
13. Patients who, in the opinion of the investigator, are not suitable for participation in this study.

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 1084 (Estimated)
Dates: Start 2023-07 (Estimated); Primary Completion 2027-06 (Estimated); Study Completion 2027-12 (Estimated)

PRIMARY OUTCOMES:
HBsAg negative conversion rate after 96 weeks of treatment | 96 weeks
  After 96 weeks of treatment, 5 ml of blood will be drawn from the patient, serum will be extracted, and HBsAg values will be quantified by chemiluminescence assay; samples less than 0.5 ng/ml will be judged as negative.
HBsAb conversion rate after 96 weeks of treatment | 96 weeks
  After 96 weeks of treatment, 5 ml of blood will be drawn from the patient, serum will be extracted, and HBsAb values will be quantified by chemiluminescence; samples greater than 10 miu/ml 0.5 will be judged as positive.

CONTACTS AND LOCATIONS:
Overall Officials: Jiabing Li, MD, Study Chair — The First Affiliated Hospital of Anhui Medical University
Locations (1):
- The First Affiliated Hospital of Anhui Medical University, Hefei, Anhui, China

IPD SHARING:
Plan to Share IPD: No